CLINICAL TRIAL: NCT00062946
Title: PET Imaging of Dopamine D2 Receptors and Extracellular Dopamine With (18F)Fallypride, D-amphetamine, and Alpha-Methyl-Para-Tyrosine in Healthy Subjects
Brief Title: PET Imaging of Dopamine in Healthy Study Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030104; 03-M-0104
Record Dates: First submitted 2003-06-17; First posted 2003-06-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-08-15

CONDITIONS: Healthy
Keywords: Thalamus; Cerebral Cortices; Quantification; Reproducibility; Dopamine Release; (18F) Fallypride; D-Amphetamine; Alpha-Methyl-Para-Tyrosine (AMPT); PET; Dopamine D2 Receptor; Healthy Volunteer; HV
MeSH Terms: interventions — N-((1-allyl-2-pyrrolidinyl)methyl)-5-(3-fluoropropyl)-2,3-dimethoxybenzamide

INTERVENTIONS:
Drug: (18F)fallypride

SUMMARY:
The purpose of this study is to measure molecules on or in cells that interact with a chemical in the nervous system, called dopamine. Investigators will obtain two kinds of images of the brain-a position emission tomography (PET) scan and a magnetic resonance imaging (MRI) scan.

Thirty-eight participants aged 18 to 45 will be enrolled in this study. They must have no history of medical or psychiatric illness, including substance abuse. Participants will have four appointments at NIH. On the first visit, they will undergo a physical exam, a medical history, and lab tests. The second and third visits will involve PET scans and the fourth visit will involve an MRI scan.

Participants will be compensated up to $430 for their involvement in this study.

DETAILED DESCRIPTION:
Abnormalities of dopaminergic function have been implicated in a number of neurological and psychiatric illnesses, including Parkinson's disease, schizophrenia, and psychostimulant dependence syndromes. Functional imaging with positron emission tomography (PET) and single photon emission computed tomography (SPECT) have demonstrated the feasibility of in vivo measurement of the distribution and the density of dopamine (DA) D1 and D2 receptors in humans. Besides simple measurement of receptor density, it has been shown that the competition between endogenous neurotransmitters and radiolabeled tracers might provide a tool to estimate extracellular levels of neurotransmitters. However, most of those studies have been confined to the striatum. In this protocol using a PET tracer (18F)fallypride, we will estimate both stimulant-induced DA release and baseline DA levels in the striatum and extrastriatal regions by comparing baseline scans and those after d-amphetamine or alpha-methyl-para-tryosine (AMPT) adminstration. In addition, to explore genetic factors that determine synaptic DA levels, allelic variations of two genes that regulate DA levels, catechol-O-methyltransferase and dopamine transporter, will be studied.

A recent study showed that oral administration of d-amphetamine induced displacement of (11C) raclopride in a similar way as the commonly used method of i.v. administration. The current protocol will be performed in two steps. First, the method of d-amphetamine administration will be determined by studying effects of oral d-amphetamine on the binding of (18F) fallypride binding. If oral administration effectively displaces the radioligand binding, this method will be applied in the subsequent study of examining effects of each of d-amphetamine and AMPT in individual subjects.

If this study successfully detects the influence of DA levels on (18F)fallypride binding, the same design will be applied to the studies of patients with psychiatric and neurological disorders.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 18-45, inclusive

In good general health on basis of history and physical examination

Normal screening laboratory studies including thyroid function tests, blood count, serum electrolytes, liver and kidney function, and urinalysis

Normal ECG at a resting condition

Normal blood pressure

No illegal drug use based on urine drug screen

EXCLUSION CRITERIA:

Pregnancy/Nursing

Evidence of active mental or neurological illness

Medically significant biochemical or hematological abnormality on screening laboratory studies

Abnormal ECG

High Blood Pressure (above 140 systolic and/or above 90 dystolic pressure)

History of myocardial infarction or angina pectoris

Positive urine drug screen or use of alcohol within one week prior to each PET study

History of substance abuse or dependence within 6 months

Presence of ferromagnetic metal in the body or heart pacemaker

Body weight more than 93 kg to limit AMPT dose to 4 g/ day (only for subjects having four PET scans and d-amphetamine and AMPT administration)

Claustrophobia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45
Dates: Start 2003-06-17; Study Completion 2007-08-15

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Anand A, Verhoeff P, Seneca N, Zoghbi SS, Seibyl JP, Charney DS, Innis RB. Brain SPECT imaging of amphetamine-induced dopamine release in euthymic bipolar disorder patients. Am J Psychiatry. 2000 Jul;157(7):1108-14. doi: 10.1176/appi.ajp.157.7.1108. PMID 10873919